CLINICAL TRIAL: NCT01739257
Title: Use of Theater to Invoke Empathy and Reduce Bias in Medical Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: The Arnold P. Gold Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 254423
Record Dates: First submitted 2012-11-26; First posted 2012-12-03 (Estimated); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Medical Student Bias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Theater (Experimental): 1-hour dramatic reading of "The Most Massive Woman Wins"
  Interventions: Behavioral: Dramatic Reading
- Lecture (Active Comparator): 1-hour lecture on the medical management of obese patients
  Interventions: Behavioral: Medical Lecture

INTERVENTIONS:
Behavioral: Medical Lecture
  Arms: Lecture
Behavioral: Dramatic Reading
  Arms: Theater

SUMMARY:
The effect of medical humanities on medical student bias and clinical management is unclear. This study characterized medical student attitudes toward obese individuals and whether reading a play employing empathic characters can modulate negative reactions.

ELIGIBILITY:
Inclusion Criteria:

* medical student at UC Davis, UC Irvine, or Mayo Medical School

Exclusion Criteria:

* none

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2012-08; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Explicit fat bias | four months
  Assessment of conscious bias against fat people (unit of measure from 11 to 99).
implicit fat bias | four months
  Measurement using the implicit association test (IAT) with scores from -2.0 to +2.0.
empathy scale | four months
  Score of Jefferson Scale of Physician Empathy (JSPE) from 20 to 180.

SECONDARY OUTCOMES:
Patient-Centered Care | four months
  Open-ended question on the clinical management of an asymptomatic, obese, elderly woman who is otherwise healthy, with coding for a response that is either patient-centered (ie: asking patient preferences and goals) or prescriptive (ie: telling the patient to diet and/or exercise).
Appraisal of obesity | four months
  An open-ended question asking participants whether they felt obesity was primarily an issue of discrimination (ie: civil rights) or a public health concern (ie: medical).

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Kravitz, MD, MSPH, Principal Investigator — UC Davis School of Medicine; Rachel Hammer, BA, Study Director — Mayo Medical School; Johanna Shapiro, PhD, Study Director — UC Irvine School of Medicine
Locations (1):
- UC Davis School of Medicine, Sacramento, California, United States